CLINICAL TRIAL: NCT03281876
Title: An Observer-blind Study to Evaluate the Efficacy, Safety, Reactogenicity and Immunogenicity of the GSK Biologicals' Investigational Vaccine GSK3277511A When Administered to COPD Patients
Brief Title: A Study to Test if the Vaccine is Working Well in Chronic Obstructive Pulmonary Disease (COPD) Patients Aged 40 to 80 Years Old to Reduce Episodes of Worsening Symptoms and to Gather Further Information on Safety and Immune Response.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 207489; 2017-000880-34 (EudraCT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-13 (Actual); Results first posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Disorders
Keywords: Immunogenicity; Vaccination; Chronic Obstructive Pulmonary Disease; Non-typeable Haemophilus influenzae; Acute exacerbation of COPD; Moraxella catarrhalis; Efficacy; Safety
MeSH Terms: conditions — Respiration Disorders; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Phase IIB, randomised, observer-blind, placebo-controlled, multi-centric study with two parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Data will be collected in an observer-blind manner. By observer-blind, it is meant that during the course of the study, the vaccine recipient and those responsible for the evaluation of any study endpoint (e.g. safety, reactogenicity and efficacy) will all be unaware of whether vaccine or placebo was administered. Each study site is responsible for having a blinding plan. To work in an observer-blind manner, vaccine preparation and administration will be done by authorised medical personnel who will not participate in any of the study clinical evaluation assays. Two teams of study personnel will hence be set up:
  * A team of unblinded personnel (responsible for the preparation and the administration of the vaccines)
  * A team of blinded personnel (responsible for the clinical evaluation of the subjects).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK3277511A Group (Experimental): Healthy males and females, 40 to 80 years of age, who received two doses of the adjuvanted GSK3277511A investigational vaccine containing surface protein D (PD), protein E- type IV pilus assembly protein (PE-PilA,) and ubiquitous surface protein A2 (UspA2) at Day 1 and Day 61.
  Interventions: Biological: NTHi Mcat investigational vaccine (GSK3277511A)
- CONTROL Group (Placebo Comparator): Healthy males and females, 40 to 80 years of age, who received two doses of placebo vaccine at Day 1 and Day 61.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: NTHi Mcat investigational vaccine (GSK3277511A) — Two doses administered intramuscularly at Day 1 and Day 61 in the deltoid region of the non-dominant arm.
  Arms: GSK3277511A Group
Biological: Placebo — Two doses administered intramuscularly at Day 1 and Day 61 in the deltoid region of the non-dominant arm.
  Arms: CONTROL Group

SUMMARY:
The purpose of this study is to test if the vaccine is working well in COPD patients aged 40 to 80 years old to reduce episodes of worsening symptoms ("exacerbations") and to gather further information on safety and immune response.

In the current study, COPD patients with a history of acute exacerbations will receive 2 doses of the investigational vaccine or placebo intramuscularly according to a 0, 2 month vaccination schedule, in addition to standard care.

The effect of vaccination against two pathogens known to cause exacerbations (Non-typeable Haemophilus influenza [NTHi] and Moraxella catarrhalis [Mcat]) will be evaluated at pre-defined timepoints (scheduled study visits).

In addition to the scheduled study visits, additional study visit(s) and/ or phone contact(s) will take place for each acute exacerbation of COPD occurring from first vaccination up to study conclusion.

DETAILED DESCRIPTION:
The purpose of this Phase IIB proof-of-concept (POC) study in moderate to very severe COPD patients (i.e. GOLD grade 2, 3 and 4) aged 40 to 80 years with a history of moderate or severe acute exacerbations of COPD (AECOPD) in the previous 12 months is to evaluate whether the NTHi-Mcat vaccine can reduce the frequency of AECOPD in this population and to assess the vaccine's safety, reactogenicity and immunogenicity.

Several formulations of a vaccine containing the NTHi antigens (low or high formulation) either non-adjuvanted or combined with different adjuvants (aluminium [Al], adjuvant system) were already evaluated in two previous Phase I clinical trials (NTHI-002 in healthy adults aged 18 - 40 years and NTHI-003 in current and former healthy smokers of 50-70 years old). The investigational vaccines were well-tolerated, with an acceptable safety and reactogenicity profile. These studies allowed the dose selection of the NTHi antigens (low formulation) and the adjuvant system currently evaluated for the first time in moderate and severe COPD patients aged 45 - 81 years in the Phase II study NTHI-004.

The safety, reactogenicity and immunogenicity of different formulations of the NTHi-Mcat investigational vaccine have been evaluated in the Phase I study in healthy adults aged 19 - 40 years and in current and former smokers aged 50 - 70 years (study NTHI MCAT-001). Based on results obtained up to 30 days post-Dose 2 from this study, the adjuvanted formulation containing NTHi proteins PD and PE-PilA and of UspA2 has been selected for evaluation in the current NTHI MCAT-002 study. Placebo will be used as a control. The NTHi-Mcat investigational vaccine and placebo will be given on top of standard of care to subjects in the respective study groups.

In the current study, moderate, severe and very severe COPD patients (i.e. GOLD grade 2, 3 and 4) with a history of AECOPD will receive 2 doses of the NTHi-Mcat investigational vaccine or placebo intramuscularly (IM) according to a 0, 2 month vaccination schedule, in addition to standard care.

Scheduled study visits, during which the effect of immunisation against NTHi and Mcat will be evaluated, will take place at pre-defined timepoints.

In addition to the scheduled study visits, ad hoc AECOPD-driven study visit(s) and/ or phone contact(s) will take place for each AECOPD occurring from first vaccination up to study conclusion:

* An AECOPD visit will be scheduled as soon as possible after the onset of the AECOPD symptoms (maximum 96 hours after the onset of the symptoms).
* Follow-up visit(s) and/or phone call(s) will take place to determine the end of the AECOPD.

Rationale for the protocol amendment:

* CD8+ T cell component was removed from the secondary endpoint, but kept in the exploratory/tertiary endpoint. Previous clinical studies have shown that the investigational NTHi and NTHi-Mcat vaccines do not induce CD8+ T cell responses. This was observed in all studies performed with the NTHi vaccine and seen in the interim analysis of NTHi Mcat-001 study.
* An exclusion criterion was updated to clarify that only subjects with clinically significant respiratory diseases other than COPD (e.g. clinically significant lung fibrosis, clinically significant pulmonary embolism) need to be excluded from study participation.
* The polymerase chain reaction (PCR) assay for sputum samples was not designed to discriminate amongst Haemophilus influenzae (Hi) serotypes. Results from AERIS epidemiological study [Wilkinson, 2017] showed that more than 99% of these bacteria would be Non-Typeable Haemophilus influenzae (NTHi). Therefore, the protocol was updated to clarify that the presence of Hi bacteria in sputum during exacerbation will be used to determine AECOPD associated to NTHi.
* The list of potential immune mediated diseases was updated (effective June 30th 2017).
* The 87% confidence interval (CI) was removed from all secondary analyses. This confidence interval will only be maintained for the primary analysis because the 95% CIs are underpowered for this study. All other sensitivity analyses on different cohorts will be described using 95% CIs. As the primary objective will have both 87% and 95%, the sensitivity analyses can be interpreted with 95% CIs.
* A Full-Analysis Set (FAS) that corresponds to an intent-to-treat analysis was added. The FAS will include all randomized subjects who will receive at least 1 vaccine administration and, as per intention-to-treat principle, a subject in the FAS will be analysed "as randomized" (i.e. according to the vaccine a subject was planned to receive irrespectively of his/her real exposure).
* Cut-off values for anti-PE, anti-PilA and anti-UspA2 antibody ELISAs were updated following the re-set up of the assays.
* Additional minor updates were based on the scientific and operational experience gained from current COPD studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* A male or female between, and including, 40 and 80 years of age at the time of the first vaccination.
* Confirmed diagnosis of COPD with forced expiratory volume in 1 second (FEV1) over forced vital capacity (FVC) ratio (FEV1/FVC) < 0.7, AND FEV1 < 80% predicted (GOLD 2, 3 and 4).
* Current or former smoker with a cigarette smoking history of ≥ 10 pack-years.
* Stable COPD patient* with documented history** of at least 1 moderate or severe AECOPD within the 12 months before Screening.

  * Patient for whom the last episode of AECOPD is resolved for at least 30 days at the time of first vaccination.

    * A documented history of a COPD exacerbation is a medical record of worsening COPD symptoms that required systemic/oral corticosteroids and/or antibiotics (for a moderate exacerbation) or hospitalization (for a severe exacerbation). Prior use of antibiotics alone does not qualify as an exacerbation history unless the use was associated with treatment of worsening symptoms of COPD, such as increased dyspnea, sputum volume, or sputum purulence. Subject verbal reports are not acceptable.
* Capable of complying with the daily electronic Diary Card completion throughout the study period, according to investigator's judgement at Visit 1.
* Female subjects of non-childbearing potential may be enrolled in the study. Non-childbearing potential is defined as pre-menarche, current bilateral tubal ligation or occlusion, hysterectomy, bilateral ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

has practiced adequate contraception for 30 days prior to vaccination, and has a negative pregnancy test on the day of vaccination, and has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the first dose of study vaccine (Day -29 to Day 1), or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Administration of immunoglobulins or any blood products within the 3 months preceding the first dose of study vaccine or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Planned administration/ administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first dose and ending 30 days after the last dose of vaccine, with the exception of any influenza or pneumococcal vaccine which may be administered ≥15 days preceding or following any study vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine dose (e.g. methotrexate).
* Administration of systemic corticosteroids within the 30 days before first vaccination.

Subjects who received systemic corticosteroids within this period may be enrolled at a later date if enrolment is still open.

Inhaled and topical steroids are allowed.

• Administration of systemic antibiotics within the 30 days before first vaccination.

Subjects who received systemic antibiotics within this period may be enrolled at a later date if enrolment is still open.

* Chronic use of antibiotics for prevention of AECOPD (e.g. azithromycin).
* Acute disease and/or fever at the time of first vaccination. Fever is defined as temperature ≥37.5°C. The preferred location for measuring temperature in this study will be the oral cavity or the axilla.

Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may be enrolled at the discretion of the investigator.

* Oxygen therapy: Use of long-term oxygen therapy (LTOT) described as resting oxygen therapy >3L/min (Oxygen use ≤3L/min flow is not exclusionary).
* Planned lung transplantation.
* Lung resection: Subjects with planned lung volume reduction surgery during the study or within the 12 months prior to first vaccination.
* Diagnosis of α-1 antitrypsin deficiency as the underlying cause of COPD.
* Diagnosed with a respiratory disorder other than COPD at time of enrolment (such as sarcoidosis, active tuberculosis, clinically significant bronchiectasis, clinically significant lung fibrosis, clinically significant pulmonary embolism, clinically significant pneumothorax, current diagnosis of asthma in the opinion of the investigator), or chest X-ray/ CT scan revealing evidence of clinically significant abnormalities not believed to be due to the presence of COPD. Subjects with allergic rhinitis do not need to be excluded and may be enrolled at the discretion of the investigator.
* History of immune-mediated disease other than COPD. If the subject has any condition on the non-exhaustive list of potential immune-mediated diseases defined in the protocol, they must be excluded unless the aetiology is clearly documented to be non-immune mediated.
* Previous vaccination with any vaccine containing NTHi and/ or Mcat antigens.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines and/ or the bronchodilator used for spirometry assessment during the study.
* Contraindication for spirometry testing.
* Unstable or life threatening cardiac disease: subjects with any of the following at Screening (Visit 1) would be excluded:

Myocardial infarction or unstable angina in the last 6 months. Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months NYHA Class IV Heart failure

* Malignancies within the previous 5 years or lymphoproliferative disorder.
* Any known disease or condition likely to cause death during the study period.
* Pregnant or lactating female.
* Current alcoholism and/or drug abuse.
* Other condition which the investigator judges may put the safety of the subject at risk through study participation or which may interfere with the study findings.
* Planned move to a location that will complicate participation in the trial through study end.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 606 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (63):
- United States (23):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Palm Springs, California
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Council Bluffs, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Mooresville, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Corvallis, Oregon
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Abingdon, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Wenatchee, Washington
- Belgium (6):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Genk
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Liège
- Canada (7):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Halifax, Nova Scotia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
- France (4):
  - GSK Investigational Site, Brest
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
- Germany (5):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Immenhausen, Hesse
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Magdeburg
- Italy (5):
  - GSK Investigational Site, Cona (FE), Emilia-Romagna
  - GSK Investigational Site, Parma, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza, Lombardy
  - GSK Investigational Site, Negrar, Veneto
- Spain (7):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Centelles (Barcelona)
  - GSK Investigational Site, Elda
  - GSK Investigational Site, La Roca Del Valles (Barcelona)
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pozuelo de Alarcón/Madrid
  - GSK Investigational Site, Vic
- United Kingdom (6):
  - GSK Investigational Site, Portsmouth, Hampshire
  - GSK Investigational Site, Bradford
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, High Heaton, Newcastle Upon Tyne
  - GSK Investigational Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Arora AK, Chinsky K, Keller C, Mayers I, Pascual-Guardia S, Vera MP, Lambert C, Lombardi S, Rondini S, Tian S, Ulloa-Montoya F, Moraschini L, Casula D; NTHi-Mcat-002 study group. A detailed analysis of possible efficacy signals of NTHi-Mcat vaccine against severe COPD exacerbations in a previously reported randomised phase 2b trial. Vaccine. 2022 Sep 29;40(41):5924-5932. doi: 10.1016/j.vaccine.2022.08.053. Epub 2022 Sep 6. PMID 36068109
- [Derived] Andreas S, Testa M, Boyer L, Brusselle G, Janssens W, Kerwin E, Papi A, Pek B, Puente-Maestu L, Saralaya D, Watz H, Wilkinson TMA, Casula D, Di Maro G, Lattanzi M, Moraschini L, Schoonbroodt S, Tasciotti A, Arora AK, Maltais F; NTHi-Mcat-002 study group. Non-typeable Haemophilus influenzae-Moraxella catarrhalis vaccine for the prevention of exacerbations in chronic obstructive pulmonary disease: a multicentre, randomised, placebo-controlled, observer-blinded, proof-of-concept, phase 2b trial. Lancet Respir Med. 2022 May;10(5):435-446. doi: 10.1016/S2213-2600(21)00502-6. Epub 2022 Jan 10. PMID 35026180

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK3277511A Group: Healthy males and females, 40 to 80 years of age, who received two doses of the adjuvanted GSK3277511A investigational vaccine containing surface protein D (PD), protein E- type IV pilus assembly protein (PE-PilA,) and ubiquitous surface protein A2 (UspA2), administered at Day 1 and Day 61
- Control Group: Healthy males and females, 40 to 80 years of age, who received two doses of placebo, administered at Day 1 and Day 61.
Period: Overall Study
Arm/Group | GSK3277511A Group | Control Group
Started | 304 | 302
Completed | 281 | 263
Not Completed | 23 | 39
Not completed — Adverse Event | 4 | 15
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 11 | 15
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 2 | 0
Not completed — OTHER | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3277511A Group | Control Group | Total
Number analyzed (Participants) | 304 | 302 | 606
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (7.5) | 66.3 (7.3) | 66.0 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 125 | 245
  Male | 184 | 177 | 361
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 0 | 1 | 1
  Asian - Central / South Asian Heritage | 2 | 0 | 2
  Asian - South East Asian Heritage | 0 | 1 | 1
  Black Or African American | 5 | 4 | 9
  Other | 1 | 0 | 1
  White - Arabic / North African Heritage | 2 | 0 | 2
  White - Caucasian / European Heritage | 294 | 296 | 590

OUTCOME MEASURES:

1. Primary Outcome: Rate of Moderate and Severe AECOPD (Any Cause)-Analysis (87% Confidence Interval [CI]), Post-dose 2 and Lasting for 1 Year
Description: Efficacy of the investigational vaccine was measured by the rate of moderate and severe AECOPD from 1-month post dose 2 up to study end (i.e. rate expressed per year and calculated as the total number of events over the follow-up exposure time). The CIs of the rate is computed using a model which accounts for repeated events. Anthonisen criteria used to detect potential AECOPD: Worsening of 2 or more of the following major symptoms for at least 2 consecutive days: dyspnoea, sputum volume, sputum purulence, OR Worsening of any major symptom together with any of the following minor symptoms for at least 2 consecutive days: sore throat, cold, fever without other cause, increased cough, increased wheeze. Moderate AECOPD requires treatment with systemic corticosteroids and/ or antibiotics. Severe AECOPD requires hospitalization. Confirmation of any AECOPD was as per investigator's judgement.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: The analysis was performed on the Modified Total Vaccinated cohort, which includes all vaccinated subjects with 2 documented study vaccine administrations with respect to the vaccine actually administered.
Measure: Number (87% Confidence Interval); unit: exacerbations per person-year
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person-year | 1.22 [1.09 to 1.36] | 1.17 [1.06 to 1.3]
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; To assess efficacy of the investigational vaccine as compared to the placebo control with respect to the rate of moderate and severe AECOPDs; Test type: Other — Vaccine Efficacy is defined as 1 minus the risk ratio (Rvacc / Rcon) based on the number of moderate and severe AECOPD observed in 1 year , with Rvacc = average yearly incidence rate of AECOPD events per subject in the GSK3277511A Group and Rcon = average yearly incidence rate of AECOPD events per subject in the Control group. The objective is to be considered a success if the lower limit of the 87% CI is above 0%; p = 0.8157, Negative Binomial regression; Negative Binomial model with arm, country, gold grade, history of exacerbation and age category as covariates and log time as offset variable; Other: Vaccine Efficacy rate = -2.26, 87% CI 2-sided [-18.27 to 11.58]

2. Primary Outcome: Rate of Moderate and Severe AECOPD (Any Cause) -Analysis (95% CI), Post-dose 2 and Lasting for 1 Year
Description: as for outcome 1
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: exacerbations per person-year
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person-year | 1.22 [1.05 to 1.41] | 1.17 [1.02 to 1.34]
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; [analysis description as in outcome 1, analysis 1]; Test type: Other — Vaccine Efficacy is defined as 1 minus the risk ratio (Rvacc / Rcon) based on the number of moderate and severe AECOPD observed in 1 year , with Rvacc = average yearly incidence rate of AECOPD events per subject in the GSK3277511A Group and Rcon = average yearly incidence rate of AECOPD events per subject in the Control group; p = 0.8157, Negative Binomial regression; [statistical method as in outcome 1, analysis 1]; Other: Vaccine Efficacy rate = -2.26, 95% CI 2-sided [-23.45 to 15.29]

3. Secondary Outcome: Number of Subjects Reported With Each Solicited Local Adverse Event (AE)
Description: Assessed solicited local symptoms were pain, redness and swelling
Time Frame: During the 7-day follow-up period (the day of vaccination + 6 days) after each vaccination administered approximately at Day 1 and Day 61
Population: The analysis was performed on the Total Vaccinated cohort which includes all vaccinated subjects with at least one documented study vaccine administration and who provided solicited safey data.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 292 | 291
Participants
  Pain, Dose 1 | 153 | 16
  Pain, Dose 2: number analyzed (Participants) | 265 | 273
  Pain, Dose 2 | 163 | 13
  Redness (mm), Dose 1 | 18 | 1
  Redness (mm), Dose 2: number analyzed (Participants) | 265 | 273
  Redness (mm), Dose 2 | 37 | 0
  Swelling (mm), Dose 1 | 13 | 2
  Swelling (mm), Dose 2: number analyzed (Participants) | 265 | 273
  Swelling (mm), Dose 2 | 31 | 0

4. Secondary Outcome: Number of Subjects Reported With Each Solicited General AE
Description: Assessed solicited general symptoms were Chills, fatigue, fever [defined as (oral cavity or axillary) temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain], headache and myalgia.
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 292 | 291
Participants
  Chills, Dose 1 | 29 | 35
  Chills, Dose 2: number analyzed (Participants) | 265 | 273
  Chills, Dose 2 | 35 | 28
  Fatigue, Dose 1 | 157 | 167
  Fatigue, Dose 2: number analyzed (Participants) | 265 | 273
  Fatigue, Dose 2 | 136 | 130
  Fever, Dose 1 | 24 | 25
  Fever, Dose 2: number analyzed (Participants) | 265 | 273
  Fever, Dose 2 | 18 | 11
  Gastrointestinal symptoms, Dose 1 | 47 | 54
  Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 265 | 273
  Gastrointestinal symptoms, Dose 2 | 39 | 35
  Headache, Dose 1 | 98 | 76
  Headache, Dose 2: number analyzed (Participants) | 265 | 273
  Headache, Dose 2 | 75 | 64
  Myalgia, Dose 1 | 78 | 72
  Myalgia, Dose 2: number analyzed (Participants) | 265 | 273
  Myalgia, Dose 2 | 74 | 43

5. Secondary Outcome: Number of Subjects Reported With Any Unsolicited Adverse Event (AE)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for any solicited symptoms.
Time Frame: During the 30-day follow-up period (the day of vaccination + 29 days) after each vaccination administered approximately at Day 1 and Day 61
Population: The analysis was performed on the Total Vaccinated cohort which includes all vaccinated subjects with at least one documented study vaccine administration and who provided unsolicited safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 304 | 302
Participants | 110 | 103

6. Secondary Outcome: Number of Subjects Reported With Any Potential Immune-mediated Diseases (pIMDs)
Description: pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From first vaccination (Day 1) up to Study end (at Day 451)
Population: The analysis was performed on the Total Vaccinated cohort which includes all vaccinated subjects with at least one documented study vaccine administration and who provided safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 304 | 302
Participants | 6 | 3

7. Secondary Outcome: Number of Subjects Reported With Any Serious Adverse Event (SAE)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity
Time Frame: From first vaccination (Day 1) up to Study end (at Day 451)
Population: The analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects with at least one documented study vaccine administration and who provided safety data.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 304 | 302
Participants | 89 | 99

8. Secondary Outcome: Rate of Moderate and Severe AECOPD in Vaccinated and Control Subjects, One Year Follow up Starting 1 Month Post Dose 2, by 3 Months Period
Description: The rates of AECOPD were expressed per year and calculated as the total number of events over the follow-up exposure time. The CIs of the rate was computed using a model which accounts for repeated events. The severity of AECOPD can be graded according to the intensity of medical intervention required. Moderate AECOPD= requires treatment with systemic corticosteroids and/or antibiotics. Severe AECOPD= requires hospitalization. The intention of the analysis of the Rate during 3, 6 and 9 months observation starting 1 month post-Dose 2 was to report the rate by 3 months period, so for the periods: 0-3, 3-6, 6-9, 9-12 months.
Time Frame: During following periods: from 0 to 3 months, from 3 to 6 months, from 6 to 9 months, from 9 to 12 months (observation starting 1 month post-Dose 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: exacerbations per person-year
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person-year
  FROM 0 TO 3 MONTHS | 1.35 [1.1 to 1.66] | 1.15 [0.92 to 1.43]
  FROM 3 TO 6 MONTHS: number analyzed (Participants) | 274 | 288
  FROM 3 TO 6 MONTHS | 1.33 [1.08 to 1.63] | 1.44 [1.19 to 1.75]
  FROM 6 TO 9 MONTHS: number analyzed (Participants) | 272 | 280
  FROM 6 TO 9 MONTHS | 1.36 [1.11 to 1.67] | 1.19 [0.96 to 1.48]
  FROM 9 TO 12 MONTHS: number analyzed (Participants) | 271 | 272
  FROM 9 TO 12 MONTHS | 0.87 [0.69 to 1.11] | 0.9 [0.71 to 1.14]

9. Secondary Outcome: Rate of Any AECOPD Case in Vaccinated and Control Subjects, One Year Follow up Starting 1 Month Post Dose 2, by 3 Months Period
Description: The rates of any AECOPD were expressed per year and calculated as the total number of events over the follow-up exposure time. The CIs of the rate was computed using a model which accounts for repeated events. The intention of the analysis of the Rate during 3, 6, 9 and 12 months observation starting 1 month post-Dose 2 was to report the rate by 3 months period, so for the periods: 0-3, 3-6, 6-9, 9-12 and 0-12 months.
Time Frame: During following periods: from 0 to 3 months, from 3 to 6 months, from 6 to 9 months, from 9 to 12 months, 0-12 months (observation starting 1 month post-Dose 2)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: exacerbations per person-year
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person-year
  FROM 0 TO 3 MONTHS | 1.47 [1.21 to 1.79] | 1.33 [1.09 to 1.63]
  FROM 3 TO 6 MONTHS: number analyzed (Participants) | 274 | 288
  FROM 3 TO 6 MONTHS | 1.56 [1.29 to 1.89] | 1.56 [1.29 to 1.88]
  FROM 6 TO 9 MONTHS: number analyzed (Participants) | 272 | 280
  FROM 6 TO 9 MONTHS | 1.49 [1.23 to 1.82] | 1.29 [1.05 to 1.59]
  FROM 9 TO 12 MONTHS: number analyzed (Participants) | 271 | 272
  FROM 9 TO 12 MONTHS | 0.98 [0.78 to 1.22] | 1.04 [0.84 to 1.3]
  From 0 TO 12 MONTHS | 1.36 [1.19 to 1.57] | 1.31 [1.15 to 1.48]
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; To assess efficacy of the investigational vaccine as compared to the placebo control with respect to the rate of AECOPDs of any severity- upto 12 months follow up period; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.7700, Negative Binomial regression; Vaccine efficacy rate = -2.72, 95% CI 2-sided [-22.95 to 14.19]

10. Secondary Outcome: Exacerbation Rate of Any AECOPD Cases, Classified by Severity, One Year Follow up Starting 1 Month Post Dose 2, by 3 Months Period
Description: The exacerbation rate of any AECOPD by severity is the average number of exacerbations for each subject: It is calculated proportionally to the follow-up time per subject and then scaled to the period considered. Mean and standard deviation of the exacerbation rate are given for each period considered. The severity of AECOPD can be graded according to the intensity of medical intervention required. Mild = can be controlled with an increase in dosage of regular medications. Moderate AECOPD= requires treatment with systemic corticosteroids and/or antibiotics. Severe AECOPD= requires hospitalization. The intention of the analysis of the Rate during 3, 6 and 9 months observation starting 1 month post-Dose 2 was to report the rate by 3 months period, so for the periods: 0-3, 3-6, 6-9, 9-12 months.
Time Frame: as for outcome 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: exacerbations per person
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person
  MILD, FROM 0 TO 3 MONTHS | 0.02 (0.15) | 0.03 (0.20)
  MILD, FROM 3 TO 6 MONTHS: number analyzed (Participants) | 274 | 288
  MILD, FROM 3 TO 6 MONTHS | 0.05 (0.24) | 0.02 (0.14)
  MILD, FROM 6 TO 9 MONTHS: number analyzed (Participants) | 272 | 280
  MILD, FROM 6 TO 9 MONTHS | 0.03 (0.19) | 0.03 (0.18)
  MILD, FROM 9 TO 12 MONTHS: number analyzed (Participants) | 271 | 272
  MILD, FROM 9 TO 12 MONTHS | 0.03 (0.17) | 0.03 (0.16)
  MODERATE, FROM 0 TO 3 MONTHS | 0.29 (0.62) | 0.23 (0.48)
  MODERATE, FROM 3 TO 6 MONTHS: number analyzed (Participants) | 274 | 288
  MODERATE, FROM 3 TO 6 MONTHS | 0.27 (0.51) | 0.3 (0.57)
  MODERATE, FROM 6 TO 9 MONTHS: number analyzed (Participants) | 272 | 280
  MODERATE, FROM 6 TO 9 MONTHS | 0.3 (0.56) | 0.25 (0.51)
  MODERATE, FROM 9 TO 12 MONTHS: number analyzed (Participants) | 271 | 272
  MODERATE, FROM 9 TO 12 MONTHS | 0.2 (0.44) | 0.17 (0.42)
  SEVERE, FROM 0 TO 3 MONTHS | 0.04 (0.24) | 0.05 (0.23)
  SEVERE, FROM 3 TO 6 MONTHS: number analyzed (Participants) | 274 | 288
  SEVERE, FROM 3 TO 6 MONTHS | 0.05 (0.22) | 0.06 (0.29)
  SEVERE, FROM 6 TO 9 MONTHS: number analyzed (Participants) | 272 | 280
  SEVERE, FROM 6 TO 9 MONTHS | 0.05 (0.29) | 0.05 (0.24)
  SEVERE, FROM 9 TO 12 MONTHS: number analyzed (Participants) | 271 | 272
  SEVERE, FROM 9 TO 12 MONTHS | 0.01 (0.11) | 0.05 (0.24)

11. Secondary Outcome: Number of Subjects With First Moderate or Severe AECOPD
Description: Number of subjects with first occurrence of moderate or severe episode of AECOPD was reported, in order to compute time to first occurrence and derive the hazard rate using Cox's proportional hazard regression model.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
Participants | 158 | 176
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; Hazard rate for moderate or severe AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.5751, Regression, Cox; Analysis using Cox proportional hazard regression including history of exacerbation, study treatment, GOLD grade and age group as covariate; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.758 to 1.166]

12. Secondary Outcome: Number of Subjects With First AECOPD of Any Severity
Description: Number of subjects with first occurrence of any episode of AECOPD of any severity was reported, in order to compute time to first occurrence and derive the hazard rate using Cox's proportional hazard regression model.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
Participants | 168 | 188
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; Hazard rate for any AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.5194, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 0.934, 95% CI 2-sided [0.758 to 1.15]

13. Secondary Outcome: Number of Subjects With First AECOPD Classified by Severity
Description: Number of subjects with first occurrence of any episode of AECOPD classified by severity was reported, in order to compute time to first occurrence and derive the hazard rate using Cox's proportional hazard regression model.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
Participants
  AFTER 1 MONTH POST DOSE 2, MILD | 27 | 27
  AFTER 1 MONTH POST DOSE 2, MODERATE | 144 | 154
  AFTER 1 MONTH POST DOSE 2, SEVERE | 30 | 41
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; Hazard rate for mild AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.8581, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.616 to 1.791]
Statistical Analysis 2: Comparison: GSK3277511A Group vs Control Group; Hazard rate for moderate AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.9634, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 0.995, 95% CI 2-sided [0.792 to 1.249]
Statistical Analysis 3: Comparison: GSK3277511A Group vs Control Group; Hazard rate for severe AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.1755, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 0.722, 95% CI 2-sided [0.45 to 1.157]

14. Secondary Outcome: Number of Days With Moderate and Severe AECOPDs
Description: The length of each AECOPD was tabulated and presented via descriptive statistics (mean, Standard Deviation) and expressed in Days.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 279 | 292
Days | 16.6 (14.29) | 15.6 (13.93)

15. Secondary Outcome: Number of Days With AECOPDs of Any Severity
Description: The length of each AECOPDs was tabulated and presented via descriptive statistics (mean, Standard Deviation).
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 279 | 292
Days | 15.9 (13.79) | 15.3 (13.51)

16. Secondary Outcome: Number of Days With AECOPDs Classified by Severity
Description: The length of each AECOPDs by severity was tabulated and presented via descriptive statistics (mean, Standard Deviation).
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 279 | 292
Days
  MILD, AFTER 1 MONTH POST DOSE 2 | 8.9 (3.56) | 12.3 (9.11)
  MODERATE, AFTER 1 MONTH POST DOSE 2 | 16.1 (13.90) | 14.5 (10.50)
  SEVERE, AFTER 1 MONTH POST DOSE 2 | 20.4 (16.78) | 21.2 (23.85)

17. Secondary Outcome: Rate of Non-Typeable Haemophilus Influenzae (NTHi)-Associated and/ or Moraxella Catarrhalis (Mcat)-Associated Moderate and Severe AECOPD
Description: The rates of AECOPD were expressed per year and calculated as the total number of events over the follow-up exposure time. The CIs of the rate was computed using a model which accounts for repeated events. Respiratory pathogens NTHi and Mcat was determined by Polymerase chain reaction (PCR) analysis in sputum samples.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: exacerbations per person-year
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person-year | 0.32 [0.25 to 0.42] | 0.32 [0.24 to 0.42]

18. Secondary Outcome: Rate of NTHi-associated and/ or Mcat-associated AECOPD of Any Severity
Description: The rates of AECOPD of any severity were expressed per year and calculated as the total number of events over the follow-up exposure time. The CIs of the rate was computed using a model which accounts for repeated events. Respiratory pathogens NTHi and Mcat was determined by polymerase chain reaction (PCR) analysis in sputum samples.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: exacerbations per person- year
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person- year | 0.39 [0.30 to 0.50] | 0.35 [0.27 to 0.45]

19. Secondary Outcome: Exacerbation Rate of Any NTHi-associated and/ or Mcat-associated AECOPD Cases, Classified by Severity
Description: The exacerbation rate of any AECOPD by severity is the average number of exacerbations for each subject: it is calculated proportionally to the follow-up time per subject, and then scaled to the period considered. Mean and standard deviation of the exacerbation rate are given for the period considered. Respiratory pathogens NTHi and Mcat was determined PCR analysis in sputum samples
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: exacerbations per person
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
exacerbations per person
  MILD, AFTER 1 MONTH POST DOSE 2 | 0.06 (0.28) | 0.03 (0.21)
  MODERATE, AFTER 1 MONTH POST DOSE 2 | 0.3 (0.67) | 0.31 (0.74)
  SEVERE, AFTER 1 MONTH POST DOSE 2 | 0.02 (0.18) | 0.01 (0.11)

20. Secondary Outcome: Number of Subjects With First Moderate or Severe NTHi-associated and/or Mcat-associated AECOPD
Description: Number of subjects with first occurrence of moderate or severe NTHI-associated and/or Mcat-associated AECOPD was reported,in order to compute time to first occurrence and derive the hazard rate using Cox's proportional hazard regression model. Respiratory pathogens NTHi and Mcat was determined PCR analysis in sputum samples.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
Participants | 62 | 62
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; Hazard rate for moderate or severe NTHi-associated and/or Mcat-associated AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.9463, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 1.038, 95% CI 2-sided [0.73 to 1.477]

21. Secondary Outcome: Number of Subjects With First NTHi-associated and/or Mcat-associated AECOPD of Any Severity
Description: Number of subjects with first occurrence of NTHI-associated and/or Mcat-associated AECOPD of any severity was reported,in order to compute time to first occurrence and derive the hazard rate using Cox's proportional hazard regression model. Respiratory pathogens NTHi and Mcat was determined PCR analysis in sputum samples.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
Participants | 70 | 67
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; Hazard rate for any NTHi-associated and/or Mcat-associated AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.6042, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 1.093, 95% CI 2-sided [0.782 to 1.528]

22. Secondary Outcome: Number of Subjects With First NTHi-associated and/or Mcat-associated AECOPD, Classified by Severity
Description: Number of subjects with first occurrence of NTHI-associated and/or Mcat-associated AECOPD classified by severity was reported, in order to compute time to first occurrence and derive the hazard rate using Cox's proportional hazard regression model. Respiratory pathogens NTHi and Mcat was determined PCR analysis in sputum samples.
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 278 | 292
Participants
  AFTER 1 MONTH POST DOSE 2, MILD | 15 | 7
  AFTER 1 MONTH POST DOSE 2, MODERATE | 58 | 59
  AFTER 1 MONTH POST DOSE 2, SEVERE | 4 | 4
Statistical Analysis 1: Comparison: GSK3277511A Group vs Control Group; Hazard rate for mild NTHi-associated and/or Mcat-associated AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.0777, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 2.243, 95% CI 2-sided [0.914 to 5.504]
Statistical Analysis 2: Comparison: GSK3277511A Group vs Control Group; Hazard rate for moderate NTHi-associated and/or Mcat-associated AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.9121, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 1.021, 95% CI 2-sided [0.71 to 1.467]
Statistical Analysis 3: Comparison: GSK3277511A Group vs Control Group; Hazard rate for severe NTHi-associated and/or Mcat-associated AECOPDs, one year follow-up starting 1 month post dose 2; Test type: Other — The dependent variable is the time to first occurrence of the event. The reference is the Placebo; p = 0.8737, Regression, Cox; [statistical method as in outcome 11, analysis 1]; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.278 to 4.502]

23. Secondary Outcome: Number of Days With Moderate and Severe NTHi-associated and Mcat-associated AECOPD
Description: The length of each NTHi associated and/or Mcat associated AECOPDs was tabulated and presented via descriptive statistics (mean, Standard Deviation).
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 279 | 292
Days | 14 (10.43) | 12.3 (5.59)

24. Secondary Outcome: Number of Days With NTHi-associated and/or Mcat-associated AECOPDs of Any Severity
Description: as for outcome 23
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 279 | 292
Days | 13.3 (9.76) | 12.1 (5.72)

25. Secondary Outcome: Number of Days With NTHi-associated and/or Mcat-associated AECOPD, Classified by Severity
Description: as for outcome 23
Time Frame: From 1-month post-Dose 2 (at Day 91) up to study end (at Day 451)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 279 | 292
Days
  AFTER 1 MONTH POST DOSE 2, MILD | 9.5 (3.54) | 9.9 (6.83)
  AFTER 1 MONTH POST DOSE 2, MODERATE | 13.8 (10.41) | 12.5 (5.62)
  AFTER 1 MONTH POST DOSE 2, SEVERE | 17.3 (11.02) | 7.5 (1.00)

26. Secondary Outcome: Anti-PD Antibody Concentrations as Measured by the Enzyme-Linked Immunosorbent Assay (ELISA)
Description: Anti-Protein D (PD) antibody concentrations as determined by ELISA, and expressed as geometric mean concentrations (GMCs) in ELISA unit per milliliter (EU/mL). For anti-PD antibodies, the cut-off of the assay is 153 ELISA Units per millilitre (EU/mL.)
Time Frame: At Day 1, Day 31, Day 61, Day 91, Day 271 and at Day 451
Population: The analysis was performed on the Per-Protocol immuno set for analysis of immunogenicity cohort which includes all vaccinated subjects who complied with the vaccination schedule and who have immunogenicity data for the specified timepoints.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL.
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 247 | 256
EU/mL.
  Day 1 | 103.7 [93.8 to 114.7] | 95.4 [86.3 to 105.4]
  Day 31: number analyzed (Participants) | 232 | 243
  Day 31 | 1048.1 [910.2 to 1206.8] | 98.2 [85.3 to 113.1]
  Day 61: number analyzed (Participants) | 239 | 253
  Day 61 | 654.6 [572.3 to 748.9] | 95.5 [83.6 to 109.1]
  Day 91: number analyzed (Participants) | 208 | 211
  Day 91 | 1521.4 [1357.6 to 1704.9] | 90.3 [80.6 to 101.3]
  Day 271: number analyzed (Participants) | 210 | 223
  Day 271 | 546 [480.3 to 620.8] | 94.8 [83.6 to 107.4]
  Day 451: number analyzed (Participants) | 221 | 216
  Day 451 | 444.1 [390.2 to 505.4] | 97.9 [85.9 to 111.5]

27. Secondary Outcome: Anti-PE Antibody Concentrations as Measured by ELISA
Description: Anti-Protein E (PE) antibody concentrations as determined by ELISA and expressed as GMCs in EU/mL For Anti-PE antibodies, the cut-off of the assay is 16 EU/mL.
Time Frame: At Day 1, Day 31, Day 61, Day 91, Day 271 and at Day 451
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL.
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 246 | 256
EU/mL.
  Day 1 | 20.9 [17.6 to 24.8] | 21.6 [18.2 to 25.7]
  Day 31: number analyzed (Participants) | 232 | 244
  Day 31 | 1108.1 [921.5 to 1332.5] | 20.7 [17.2 to 24.9]
  Day 61: number analyzed (Participants) | 239 | 251
  Day 61 | 872.8 [726.6 to 1048.3] | 20.5 [17.1 to 24.6]
  Day 91: number analyzed (Participants) | 208 | 211
  Day 91 | 6020 [5181.2 to 6994.7] | 20.1 [17.3 to 23.4]
  Day 271: number analyzed (Participants) | 210 | 223
  Day 271 | 1254.9 [1069.5 to 1472.5] | 19.3 [16.5 to 22.5]
  Day 451: number analyzed (Participants) | 221 | 215
  Day 451 | 835.2 [715.0 to 975.6] | 19.7 [16.8 to 23.0]

28. Secondary Outcome: Anti-PilA Antibody Concentrations as Measured by ELISA
Description: Anti-Type IV pilus assembly protein (PilA) antibody concentrations as determined by ELISA, and expressed as GMCs in EU/mL. For Anti-PilA antibodies, the cut-off of the assay is 8 EU/mL.
Time Frame: At Day 1, Day 31, Day 61, Day 91, Day 271 and at Day 451
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL.
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 247 | 256
EU/mL.
  Day 1 | 8.3 [6.9 to 9.8] | 8.5 [7.1 to 10.1]
  Day 31: number analyzed (Participants) | 231 | 243
  Day 31 | 153 [124.2 to 188.6] | 9.2 [7.5 to 11.4]
  Day 61: number analyzed (Participants) | 238 | 251
  Day 61 | 134.2 [109.7 to 164.2] | 8.8 [7.2 to 10.8]
  Day 91: number analyzed (Participants) | 208 | 211
  Day 91 | 913.5 [770.5 to 1082.9] | 8.9 [7.5 to 10.5]
  Day 271: number analyzed (Participants) | 210 | 223
  Day 271 | 189.6 [159.2 to 225.7] | 8 [6.8 to 9.5]
  Day 451: number analyzed (Participants) | 221 | 216
  Day 451 | 126.5 [106.1 to 150.8] | 8.3 [6.9 to 9.9]

29. Secondary Outcome: Anti-UspA2 Antibody Concentrations as Measured by ELISA
Description: Anti-ubiquitous surface protein A2 of Moraxella catarrhalis (UspA2) aantibody concentrations as determined by ELISA, and expressed as GMCs in EU/mL. For Anti-UspA2 antibodies, the cut-off of the assay is 28 EU/mL.
Time Frame: At Day 1, Day 31, Day 61, Day 91, Day 271 and at Day 451
Population: as for outcome 26
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 246 | 255
EU/mL
  Day 1 | 540.3 [452.6 to 645.0] | 604.7 [507.2 to 721.0]
  Day 31: number analyzed (Participants) | 232 | 242
  Day 31 | 1092.1 [997.5 to 1195.5] | 485.2 [442.9 to 531.6]
  Day 61: number analyzed (Participants) | 238 | 251
  Day 61 | 848.7 [781.5 to 921.5] | 473.5 [436.2 to 513.9]
  Day 91: number analyzed (Participants) | 208 | 211
  Day 91 | 1223.7 [1110.8 to 1348.0] | 446 [404.5 to 491.8]
  Day 271: number analyzed (Participants) | 210 | 222
  Day 271 | 645.1 [582.1 to 714.8] | 445.4 [402.7 to 492.6]
  Day 451: number analyzed (Participants) | 221 | 215
  Day 451 | 575.9 [512.9 to 646.7] | 468.5 [416.5 to 527.1]

30. Secondary Outcome: Frequency of PD Specific Cluster of Differentiation (CD)4+ T-cells Expressing at Least 2 Markers Among CD40L, IL2, TNF-Alpha, IFN-Gamma, IL-13 and IL-17 Using Background Reduced Frequency Data
Description: The ICS staining assay was used to assess cell-mediated immunogenicity (CMI) responses. After Peripheral blood mononuclear cell (PBMC) stimulation with the relevant antigen, the frequency of PD specific CD4+ T-cells expressing selected combination of cytokines such as interleukine-2, 13, 17 (IL-2, IL-13, IL-17), interferon-gamma (IFN-γ), tumour necrosis factor-alpha (TNF-α) and cluster of differentiation 40 ligand (CD40L) are evaluated by flow cytometry and expressed as mean and standard deviation.
Time Frame: At Day 1, Day 91, Day 271 and at Day 451
Population: The analysis was performed on the Per-Protocol CMI set for analysis of immunogenicity cohort which includes all vaccinated subjects who were complied with the vaccination schedule and who have CMI data for the specified timepoints.
Measure: Mean (Standard Deviation); unit: T cells/million cells
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 47 | 41
T cells/million cells
  Day 1 | 56.6 (125.7) | 59.7 (118.2)
  Day 91: number analyzed (Participants) | 42 | 36
  Day 91 | 890.2 (988.8) | 55.8 (88.2)
  Day 271: number analyzed (Participants) | 42 | 41
  Day 271 | 364.6 (363.9) | 51.8 (90.9)
  Day 451: number analyzed (Participants) | 42 | 36
  Day 451 | 267 (282.6) | 46.7 (101.1)

31. Secondary Outcome: Frequency of PE Specific (CD)4+ T-cells Expressing at Least 2 Markers Among CD40L, IL2, TNF-Alpha, IFN-Gamma, IL-13 and IL-17 Using Background Reduced Frequency Data
Description: The ICS staining assay was used to assess CMI responses. After PBMC stimulation with the relevant antigen, the frequency of PE specific CD4+ T-cells expressing selected combination of cytokines such as (IL-2, IL-13, IL-17), IFN-γ, TNF-α and CD40L are evaluated by flow cytometry and expressed as mean and standard deviation.
Time Frame: At Day 1, Day 91, Day 271 and at Day 451
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: T cells/million cells
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 47 | 41
T cells/million cells
  Day 1 | 63.1 (211.4) | 92.9 (266.0)
  Day 91: number analyzed (Participants) | 42 | 36
  Day 91 | 797 (1082.9) | 76.2 (195.0)
  Day 271: number analyzed (Participants) | 42 | 41
  Day 271 | 384.8 (539.9) | 61.4 (207.2)
  Day 451: number analyzed (Participants) | 42 | 36
  Day 451 | 335.7 (493.7) | 81.2 (258.9)

32. Secondary Outcome: Frequency of PilA Specific CD4+ T-cells Expressing at Least 2 Markers Among CD40L, IL2, TNF-Alpha, IFN-Gamma, IL-13 and IL-17 Using Background Reduced Frequency Data
Description: The ICS staining assay was used to assess CMI responses. After PBMC stimulation with the relevant antigen, the frequency of PilA specific CD4+ T-cells expressing selected combination of cytokines such as IL-2, IL-13, IL-17, IFN-γ, TNF-α and CD40L are evaluated by flow cytometry and expressed as mean and standard deviation.
Time Frame: At Day 1, Day 91, Day 271 and at Day 451
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: T cells/million cells
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 47 | 41
T cells/million cells
  Day 1: number analyzed (Participants) | 47 | 40
  Day 1 | 26.2 (45.4) | 53.3 (95.9)
  Day 91: number analyzed (Participants) | 42 | 36
  Day 91 | 305.8 (321.7) | 44.6 (114.8)
  Day 271: number analyzed (Participants) | 42 | 41
  Day 271 | 137.3 (163.2) | 42.1 (78.2)
  Day 451: number analyzed (Participants) | 42 | 36
  Day 451 | 141 (147.1) | 42.4 (95.3)

33. Secondary Outcome: Frequency of UspA2 Specific CD4 + T-cells Expressing at Least 2 Markers Among CD40L, IL2, TNF-Alpha, IFN-Gamma, IL-13 and IL-17 Using Background Reduced Frequency Data
Description: The ICS staining assay was used to assess CMI responses. After PBMC stimulation with the relevant antigen, the frequency of UspA2 specific CD4+ T-cells expressing selected combination of cytokines such as IL-2, IL-13, IL-17, IFN-γ, TNF-α and CD40L are evaluated by flow cytometry and expressed as mean and standard deviation.
Time Frame: At Day 1, Day 91, Day 271 and at Day 451
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: T cells/million cells
Arm/Group | GSK3277511A Group | Control Group
Number analyzed (Participants) | 47 | 41
T cells/million cells
  Day 1: number analyzed (Participants) | 47 | 40
  Day 1 | 66.1 (177.1) | 47.2 (85.8)
  Day 91: number analyzed (Participants) | 42 | 36
  Day 91 | 646.3 (545.2) | 70.3 (94.6)
  Day 271: number analyzed (Participants) | 42 | 41
  Day 271 | 330.5 (278.5) | 60.8 (80.0)
  Day 451: number analyzed (Participants) | 42 | 35
  Day 451 | 331.3 (310.4) | 61.5 (89.2)

ADVERSE EVENTS:
Time Frame: Solicited AEs reported during the 7-day follow-up period and Unsolicited AEs reported during the 30-day follow-up period after any vaccination. SAEs reported from first vaccination (Day 1) up to Study end (at Day 451 - an average of 15 months).
Arm/Group | GSK3277511A Group | Control Group
All-Cause Mortality (participants affected / at risk) | 1/304 | 10/302
Serious Adverse Events (participants affected / at risk) | 89/304 | 99/302
Other Adverse Events (participants affected / at risk) | 276/304 | 247/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3277511A Group (N=304) | Control Group (N=302)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 4 (5) | 2 (2)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (3)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyschezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cirrhosis alcoholic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
CNS ventriculitis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Graft infection (Infections and infestations) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1) | 4 (5)
Influenza (Infections and infestations) | 4 (4) | 2 (2)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 15 (17)
Pneumonia pneumococcal (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Tracheobronchitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3)
Urosepsis (Infections and infestations) | 0 (0) | 2 (3)
Wound abscess (Infections and infestations) | 0 (0) | 1 (1)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anastomotic complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Drain site complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Musculoskeletal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypopharyngeal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Penile cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ruptured cerebral aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 3 (3) | 0 (0)
Device loosening (Product Issues) | 0 (0) | 1 (1)
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 7 (7)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 41 (55) | 53 (83)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4)
Aortic aneurysm (Vascular disorders) | 1 (1) | 1 (1)
Femoral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vein occlusion (Vascular disorders) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3277511A Group (N=304) | Control Group (N=302)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Dermatochalasis (Eye disorders) | 1 (1) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Retinoschisis (Eye disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 9 (9)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 71 (86) | 77 (90)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Pancreatic disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 2 (2)
Chills (General disorders) | 52 (64) | 52 (65)
Drug intolerance (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 195 (297) | 197 (299)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 43 (55) | 1 (1)
Injection site pain (General disorders) | 213 (324) | 30 (31)
Injection site reaction (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 35 (45) | 3 (3)
Malaise (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 5 (5) | 0 (0)
Pyrexia (General disorders) | 39 (42) | 32 (36)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Chronic sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 3 (3) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 2 (2)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 13 (13) | 13 (15)
Oral candidiasis (Infections and infestations) | 2 (2) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Sweat gland infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1) | 4 (5)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 115 (153) | 94 (116)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 127 (178) | 111 (145)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Post polio syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1)
Chromaturia (Renal and urinary disorders) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 1 (1)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dandruff (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral venous disease (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/76/NCT03281876/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-29): https://cdn.clinicaltrials.gov/large-docs/76/NCT03281876/SAP_001.pdf